CLINICAL TRIAL: NCT01176435
Title: Clinical Trial to Evaluate Levodopa as Treatment to Improve Vision in Individuals With Albinism
Brief Title: Trial of L-DOPA as a Treatment to Improve Vision in Albinism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0912M75653
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Results first posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Albinism
Keywords: Levodopa; Albinism; Vision
MeSH Terms: conditions — Albinism | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.76 mg/kg L-DOPA (Active Comparator): Solution taken orally three times a day.
  Interventions: Drug: Levodopa
- 0.51 mg/kg L-DOPA (Active Comparator): Solution taken orally three times a day.
  Interventions: Drug: Levodopa
- Placebo (Placebo Comparator): Solution taken orally three times a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levodopa — Solution taken orally three times a day.
  Arms: 0.76 mg/kg L-DOPA
Drug: Levodopa — Solution taken orally three times a day.
  Arms: 0.51 mg/kg L-DOPA
Drug: Placebo — Solution taken orally three times a day.
  Arms: Placebo

SUMMARY:
This project will evaluate the effect of two doses of levodopa (L-DOPA) in a randomized, placebo-controlled, double-masked clinical trial to see if vision can be improved in individuals with albinism. The hypothesis is that providing L-DOPA to the retinas of these individuals may increase melanin pigment production. Increased melanin has previously been shown to be associated with improved vision.

DETAILED DESCRIPTION:
A group of 45 individuals with the clinical findings of oculocutaneous albinism (OCA) will be randomly assigned to one of 3 treatment groups: treatment with 0.76 mg/kg/d with 25% carbidopa, 0.51 mg/kg/d levodopa with 25% carbidopa [divided into 3 doses/d), or placebo. Subjects will be between ages 3 and 60 years. Blood will be drawn to determine the mutation(s) in the genes that causes OCA. Primary outcome will be binocular best-corrected visual acuity measured with the EVA. Enrollment and 20 week examination will be complete eye exam with fundus photos. At weeks 5, 10, and 15, exams will include just vital signs and BCVA. At all visits, a review of potential side effects will be conducted. Between visits, subjects will be contacted to determine if any side effects have occurred. The study will remain double masked until the last study examination on the last subject has been performed. At that time, the data will be statistically analyzed and subjects will be informed re: treatment assignment, mutations found, and the study results.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 60 years with albinism

Exclusion Criteria:

* Glaucoma or at increased risk of glaucoma
* History of dystonia
* History of melanoma
* Planning to undergo eye muscle surgery during study time frame
* Undergoing vision therapy
* Taking iron supplements or vitamins with iron
* Taking medication for ADHD
* Known liver or gastrointestinal disease
* Previous treatment with levodopa
* Psychological problems
* Ocular abnormalities other than those associated with albinism
* Pregnant, nursing or planning to become pregnant during study
* Known allergy to levodopa/carbidopa

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Summers, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Eye Clinic, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Solution taken orally three times a day.
  Levodopa: Solution taken orally three times a day.
Period: Overall Study
Arm/Group | 0.76 mg/kg L-DOPA | 0.51 mg/kg L-DOPA | Placebo
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.76 mg/kg L-DOPA | 0.51 mg/kg L-DOPA | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Full Range); unit: years] | 12.5 [3.5 to 57] | 19.7 [4 to 49.3] | 10.6 [4 to 18.1] | 14.5 [3.5 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 5 | 24
  Male | 4 | 7 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 13 | 14 | 12 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Improved Vision
Description: Binocular best-corrected visual acuity-The visual acuity test is used to determine the smallest letters you can read on a standardized chart (Snellen chart) or a card held 20 feet (6 meters) away. Special charts are used when testing at distances shorter than 20 feet (6 meters). Ranges are 20/10 vision to 20/200 vision. 20/10 being the best and 20/200 being the worse.
Time Frame: 20 weeks
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | 0.76 mg/kg L-DOPA | 0.51 mg/kg L-DOPA | Placebo
Number analyzed (Participants) | 15 | 15 | 15
logMAR | 0.67 [0.20 to 1.0] | 0.55 [0.20 to 0.88] | 0.53 [0.20 to 0.90]

ADVERSE EVENTS:
Arm/Group | 0.76 mg/kg L-DOPA | 0.51 mg/kg L-DOPA | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 7/15 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.76 mg/kg L-DOPA (N=15) | 0.51 mg/kg L-DOPA (N=15) | Placebo (N=15)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Loss of Appetite (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dizzy when standing quickly (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Sleepiness (General disorders) | 1 (1) | 1 (1) | 1 (1)
Thirsty (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1)
Swelling of hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Twitch/Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No